CLINICAL TRIAL: NCT04369612
Title: Home Based Monitoring of Kidney Transplants Utilizing Capillary Microsamples
Acronym: HBM-KTx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anders Åsberg, Head of Laboratory, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 134787
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Kidney Transplant Failure and Rejection
Keywords: capillary sample, finger-prick, home-based monitoring
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Intervention Model Description: Two Groups, randomized 1:1, to a) Standard of care and b) home-based monitoring. Followed between 1-2 to 7-8 weeks after transplantation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Standard follow-up after kidney transplantation during the first 7-8 post-transplant weeks
  Interventions: Procedure: Standard follow-up
- Home-based monitoring (Experimental): Every second visit will be performed without patients actually visiting the hospital. They take a capillary blood sample themselves, send it to the lab and get a telecom follow-up by treating physician the same day.
  Interventions: Procedure: Home-based monitoring

INTERVENTIONS:
Procedure: Standard follow-up — Standard post-transplant follow-up
  Arms: Standard of care
Procedure: Home-based monitoring — Patients take capillary blood sample by finger-prick and send to lab for analyses. Telecom follow-up that day by treating physician
  Arms: Home-based monitoring

SUMMARY:
Renal transplant recipients are followed as out patients at the transplant center for about 8 weeks after surgery. Between 1-2 weeks after surgery, 50 standard immunological patients will be randomized (1:1) to either follow standard of care (SOC) or having every second poli clinical visit without entering the hospital HBM; Home Based Monitoring). They are to take a capillary finger-prick blood sample themselves, send it to the laboratory for analysis and then they will get a telecom follow-up that day from their transplant physician. Outcome is no difference with regards to being able to follow the randomized follow-up procedure.

DETAILED DESCRIPTION:
Renal transplant recipients are followed as out patients at the transplant center for about 8 weeks after surgery. Between 1-2 weeks after surgery, 50 standard immunological patients (i.e. first, kidney (only) transplants, no donors specific antibodies (DSA), panel reactive antibodies (PRA), ABO blood type compatible transplant) will be randomized (1:1) to either follow standard of care (SOC) or having every second poli clinical visit without entering the hospital HBM; Home Based Monitoring). They are to take a capillary finger-prick blood sample themselves and send it to the laboratory for analysis (creatinine, hemoglobin, tacrolimus and mycophenolate) and then they will get a telecom follow-up that day from their transplant physician. Outcome is no difference with regards to being able to follow the randomized follow-up procedure without having acute rejection episodes and no need for extra ou-patients visits for any reason. End of study is week 7-8 after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Kidney only transplant
* Immunosuppressive therapy With at least one of; tacrolimus, cyclosporine, everolimus, sirolimus, mycophenolate
* Standard immunological risk; no DSA, no PRA, not ABO-incompatible transplant
* Age above 18 years
* Followed at Oslo University Hospital-Rikshospitalet transplant center
* Written informed consent

Exclusion Criteria:

* Pregnant or breast feeding female recipients
* Ongoing acute rejection episodes at time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Success rate | 1-8 weeks post-transplant
  Complete follow-up without acute rejection and no need for extra visit of any cause

SECONDARY OUTCOMES:
Extra visits to Control immunosuppressive drug levels | 1-8 weeks post-transplant
  Number of extra visits in order to monitoring appropriate drug Levels of immunosuppressive drugs

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Midtvedt, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo Univeristy Hospital - Rikshospitralet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Not allowed without specific ethical committee approval